CLINICAL TRIAL: NCT00913250
Title: A Randomized, Single-Blind, Crossover Study in Healthy Volunteers to Demonstrate the Bioequivalence of AVONEX® (Interferon Beta-1a) Solutions for Injection Produced by a Serum-Containing Manufacturing Process and by a Serum-Free Manufacturing Process
Brief Title: A Bioequivalence Study of Serum Free Avonex and Serum Containing Avonex in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: C-869
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Serum containing Avonex followed by serum free Avonex
  Interventions: Drug: Serum containing Avonex
- Sequence 2 (Experimental): Serum free Avonex followed by serum containing Avonex
  Interventions: Drug: Serum Free Avonex

INTERVENTIONS:
Drug: Serum containing Avonex — 60mcg IM dose of serum containing Avonex on Day 1, followed by 60mcg IM dose of serum free Avonex on Day 15
  Other Names: Avonex
  Arms: Sequence 1
Drug: Serum Free Avonex — 60mcg IM dose of serum free Avonex on Day 1, followed by 60mcg IM dose of serum containing Avonex on Day 15.
  Other Names: Avonex
  Arms: Sequence 2

SUMMARY:
Demonstrate the bioequivalence of a serum-free solution to a serum containing solution of Avonex.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions
* History of hypersensitivity to acetaminophen (paracetamol), ibuprofen, or codeine.
* Known allergy to dry natural rubber
* History of seizure disorder or unexplained blackouts
* History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease

Other inclusion and exclusion criteria apply as per protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2003-08; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate the bioequivalence of a serum-free Avonex and a serum-containing AVONEX® when given intramuscularly (IM) to healthy volunteers. | Study duration is 72 days

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — Biogen